CLINICAL TRIAL: NCT02932995
Title: Evaluation of DUAL Drug-eluting Stent ( DXR Stent) for Vascular Healing and Thrombus Formation : an Optical Coherence Tomography Study
Brief Title: DXR Stent for Vascular Healing and Thrombus Formation: OCT Study
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Chung-Ang University (Other)
Collaborators: Konyang University Hospital (Other); Kyunghee University Medical Center (Other); Korea University Guro Hospital (Other); Ulsan University Hospital (Other); Jeju National University Hospital (Other)
Responsible Party: Principal Investigator, Sang-Wook Kim, Professor, Chung-Ang University
Other Study IDs: C2015201
Record Dates: First submitted 2016-10-12; First posted 2016-10-14 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Coronary Artery Disease; Coronary Stent Occlusion
Keywords: Optical Coherence Tomography; Drug-Eluting Stent
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- DXR stent group: Patients who undergo coronary intervention with DXR stent

SUMMARY:
The purpose of this study is to evaluate the efficacy of a novel dual drug-eluting stent (DXR stent), which slowly releases both cilostazol and paclitaxel, for strut coverage, malapposition, and thrombus formation, assessed by an optical coherence tomography.

ELIGIBILITY:
Inclusion Criteria:

1. Patient

   * Age >=19 years
   * Clinically indicated to invasive coronary angiography
   * Patient capable and willing of giving written informed consent
2. Angiographic

   * coronary artery disease confined to native coronary artery
   * >50% diameter stenosis by invasive coronary angiography
   * reference diameter 2.5-4.0mm, lesion length ≤30 mm

Exclusion Criteria:

1. Patient

   * Inability to provide written informed consent
   * Serious comorbidity which may affect the trial by decision of investigators
   * Prior CABG to target vessel
   * Congestive heart failure with NYHA Class III or IV or left ventricular ejection fraction less than 30%
   * Prior ST elevation myocardial infarction within 72 hours from the procedure
   * Hemodynamic or electrical instability including shock
   * Serious coronary artery spasm, unrelated to catheter
   * Pregnancy or possible pregnant status
   * Allergy to iodinated contrast agent
   * Serum creatinine >=1.7 mg/dL or creatinine clearance <= 30 ml/min
   * ST elevation myocardial infarction
2. Angiographic (OCT)

   * Left main disease
   * Severely calcified lesion
   * Severely tortuous, or TIMI flow grade 0 or 1 by angiography, or inappropriate for OCT procedure by investigators' decision

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who undergo coronary artery intervention with DXR stent
Sampling Method: Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-10 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Stent strut coverage (Incidence of uncovered strut) | 6 month
  Coronary angiography with OCT follow up

SECONDARY OUTCOMES:
Stent malapposition | 6 month
  Coronary angiography with OCT follow up
Stent thrombosis | 6 month
  Coronary angiography with OCT follow up

OTHER OUTCOMES:
major adverse cardiovascular event (all-cause death, stroke, unexpected revascularization) | 1 year
  Clinical outcome follow up
long term major cardiovascular event major adverse cardiovascular event (all-cause death, stroke, unexpected revascularization) | 3 year
  Clinical outcome follow up

CONTACTS AND LOCATIONS:
Overall Officials: Sang-Wook Kim, MD, PhD, Principal Investigator — Chung-Ang University Hosptial, Chung-Ang University College of Medicine
Locations (6):
- South Korea (6):
  - Konyang University Hospital, Daejeon
  - Jeju National University Hospital, Jeju City
  - KyungHee University Medical Center, Seoul
  - Chung-Ang University Hospital, Seoul
  - Korea University Guro Hospital, Seoul
  - Ulsan university hospital, Ulsan

IPD SHARING:
Plan to Share IPD: No